CLINICAL TRIAL: NCT02293421
Title: Evaluation of the STOP-BANG Screening Questionnaire in a Sleep Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Umeå University (Other); Uppsala University Hospital (Other); Stockholm Heart Center, Sweden (Unknown); Sunderbyn Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSA STOP-BANG
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STOP BANG (Other): STOP BANG screening questionnaire and a snore question
  Interventions: Other: Obstructive sleep apnea

INTERVENTIONS:
Other: Obstructive sleep apnea

SUMMARY:
Although obstructive sleep apnea (OSA) is common, most of the patients are undiagnosed. OSA is associated with a large number of co-morbidities, and thus, it is of great importance to identify the patients and start treatment in order to reduce the risks for complications. Current screening tools are quite unspecific and the golden standard methodology for diagnosis, polysomnography, is expensive and time consuming, thus not suitable for screening. In perioperative medicine the STOP BANG screening questionnaire is currently the recomended screening tool, however this questionnaire has only been evaluated in a sleep clinic in a very limited numbers of patients.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* First or part of the first visit to a sleep clinic
* Planned or just conducted polysomography

Exclusion Criteria:

* Not able to understand the information and sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
STOP BANG | At diagnosis, one time
Snore question | At diagnosis, one time
Polygraphy | At diganosis, one time
  Apnea hypopnea index (AHI, oxygen desatuaration index (ODI)

SECONDARY OUTCOMES:
Pulseoximetry | At dignosis, one time

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Anesthesiology, Surgical Sciences and Intensive Care Medicine, Karolinska University Hospital, Solna, Stockholm, Sweden

REFERENCES:
- [Derived] Christensson E, Franklin KA, Sahlin C, Palm A, Ulfberg J, Eriksson LI, Lindberg E, Hagel E, Jonsson Fagerlund M. Can STOP-Bang and Pulse Oximetry Detect and Exclude Obstructive Sleep Apnea? Anesth Analg. 2018 Sep;127(3):736-743. doi: 10.1213/ANE.0000000000003607. PMID 29958223